CLINICAL TRIAL: NCT04467749
Title: Effects of In-wheel Suspension in Reducing Vibration, Neck, and Back Pain
Brief Title: Effects of In-Wheel Suspension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Alicia Koontz, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20020199
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Spinal Cord Injuries; Fatigue; Back Pain; Neck Pain
MeSH Terms: conditions — Spinal Cord Injuries; Fatigue; Back Pain; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspension Wheel (Experimental): Participants will be given a set of in-wheel suspension wheels to use in their normal daily routine for three months.
  Interventions: Other: Suspension Wheel

INTERVENTIONS:
Other: Suspension Wheel — Participants will be given a pair of Spinergy or Loopwheels to use during the 12-week intervention period. The Spinergy wheels consist of a lightweight carbon fiber material with natural shock absorbing properties. Loopwheels offer a rigid rim, a mid-wheel shock absorbing hub and three in-wheel loops that work as a self-correcting system when encountering uneven ground.
  Other Names: Spinergy or Loopwheel

SUMMARY:
Manual wheelchairs allow individuals with spinal cord injuries (SCI) to safely and effectively access their environment. However, continual exposure to whole body vibration (WBV) is one of many contributing factors to neck pain, back pain, and fatigue in wheelchair users with SCI.

Vibration-reducing in-wheel suspension has the potential to mitigate issues associated with long-term manual wheelchair propulsion. Evidence is lacking on how well these systems work for reducing harmful shock and vibration, pain and fatigue. The purpose of this study is to examine how these wheels change the vibration levels manual wheelchair users are exposed to and how they impact pain and fatigue.

DETAILED DESCRIPTION:
Objective: The purpose of this project is to examine how Integral or in-wheel suspension impacts shock, vibration, pain and fatigue in manual wheelchair users with spinal cord injury who have chronic neck or back pain, defined as continuous or daily recurring pain that has been present for more than 3 months.

Experimental Design: This study consists of 2 phases. The first phase is a non-experimental post-test only design. The second phase is a non-experimental pretest-post-test design.

Methods: Thirty participants will be recruited to participate.

At Baseline (visit 1) participants will be asked to complete the study questionnaires and a standardized mobility course using a pair of standard wheelchair wheels (spoked rim), Spinergy lightweight carbon fiber wheels, and Loopwheels. Vibration exposure will be measured during the various propulsion tasks. The participant will be blinded to the type of wheel being used in the trial. Participants will be given a set of wheels (either Spinergy or Loopwheels) to use at home for the 12-week intervention.

Participants will use the in-wheel suspension wheels in their normal daily routine for 12-weeks. During this time, they will receive online surveys three times per week covering pain and fatigue experienced in various parts of the body.

At Closeout (Visit 2), participants will be asked to return to the lab to collect final outcomes, complete an exit survey and have their wheels swapped out for their original set.

ELIGIBILITY:
Inclusion Criteria:

* have neurological impairment secondary to a traumatic SCI
* have a SCI which occurred or was diagnosed over one year prior to the start of the study
* uses a manual wheelchair as a primary means of mobility (at least 30 hours per week but not necessarily always in motion)
* uses a manual wheelchair with 24- or 25-inch quick release wheels
* uses a manual wheelchair that does not have suspension elements in the frame,
* weighs under 265 pounds (maximum weight limit of the suspension wheels),
* has moderate chronic neck and/or back pain.
* proficient in English

Exclusion Criteria:

* History of fractures or dislocations in the shoulder, elbow and wrist from which the participant has not fully recovered (i.e. the participant may no longer experience pain or limited/altered function due to the injury)
* upper limb pain that interferes with the ability to propel,
* severe cognitive limitations,
* current or recent (within the last 6 months) history of pressure sores.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Vibrational Dose Value (VDV) | Baseline Visit (Phase 1 Primary Outcome)
  Amount of whole body vibration exposure in units of meters/sec to power of 1.75) computed using a 3-axis accelerometer attached to wheelchair on the obstacle course.
Changes in Neck Pain | Baseline and 12-weeks (Phase 2 Primary Outcome)
  Measured using the Numerical Rating Scale (NRS). The NRS measures amount of pain experienced in a body part over the last 24 hours on a scale of 0 = no pain to 10 = pain as bad as you can imagine.
Changes in Upper Back Pain | Baseline and 12-weeks (Phase 2 Primary Outcome)
  Measured using the Numerical Rating Scale (NRS). The NRS measures amount of pain experienced in a body part over the last 24 hours on a scale of 0 = no pain to 10 = pain as bad as you can imagine.
Changes in Fatigue | Baseline and 12-weeks (Phase 2 Primary Outcome)
  Measured using the Daily Questionnaire for Pain and Fatigue. Four questions ask specifically about fatigue experienced when using the wheelchair in and outside of the home and on smooth and uneven surfaces. The scale ranges from 0 = no fatigue to 3 = extreme fatigue.

SECONDARY OUTCOMES:
Changes in Mobility Participation in the Community | Baseline and 12-weeks (Phase 2 Secondary Outcome)
  Measured using Environmental Aspects of Mobility Questionnaire (EAMQ) a 36-item questionnaire accessing frequency of encounters and avoidances to environmental features. Each feature is scored on a 5-point scale (1=never, 2 = rarely, 3 = sometimes, 4=often, 5 = always). A separate total score is determined for Encounters ranging from 21 (never encounters any feature) to 105 (always encounters all features) and Avoidances ranging from 15 (never avoids any feature) to 75 (always avoids all features).

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Koontz, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in a publication related to this study, after deidentification may be shared. Requesters will be asked to submit aims and a methodologically sound proposal for which they plan to use the data to be evaluated by study team before releasing the information. The request and proposal will be directed to the corresponding author of the publication. Data requesters will also need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Data will be immediately available post acceptance date of the study related publication and for a period of 5 years.
Access Criteria: Requesters must provide methodologically sound aims and proposal describing use of the data. They also need to sign a data access agreement.